CLINICAL TRIAL: NCT06665711
Title: COMPARISON BETWEEN 3% HYPERTONIC SALINE VERSUS SALBUTAMOL IN CHILDREN WITH BRONCHIOLITIS
Brief Title: Comparison of 3% Hypertonic Saline and Salbutamol in Children With Bronchiolitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Qasim Niaz, Post Graduate Resident Pediatrics, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp125
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: BRONCHIOLITIS
Keywords: BRONCHIOLITIS
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; Albuterol

STUDY DESIGN:
Intervention Model Description: This study will employ a randomized controlled trial (RCT) design, which is considered the gold standard for evaluating the efficacy of interventions. The primary aim is to compare the effectiveness of 3% hypertonic saline against Salbutamol (Ventolin) in treating bronchiolitis in children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: 3% Hypertonic Saline (Active Comparator): In this arm of the study, participants will receive nebulized 3% hypertonic saline as the primary treatment for bronchiolitis. The administration of hypertonic saline is aimed at reducing airway edema and improving mucociliary clearance in infants experiencing respiratory distress due to bronchiolitis.
  Interventions: Procedure: 3% Hypertonic Saline
- Intervention: Salbutamol (Ventolin) (Active Comparator): In this arm of the study, participants will receive nebulized Salbutamol, a bronchodilator commonly used in the management of bronchospasm associated with respiratory conditions, including bronchiolitis. The objective is to evaluate the effectiveness of Salbutamol in comparison to 3% hypertonic saline in improving the clinical outcomes of infants with bronchiolitis.
  Interventions: Procedure: Intervention: Salbutamol (Ventolin)

INTERVENTIONS:
Procedure: 3% Hypertonic Saline — In this arm of the study, participants will receive nebulized 3% hypertonic saline as the primary treatment for bronchiolitis. The administration of hypertonic saline is aimed at reducing airway edema and improving mucociliary clearance in infants experiencing respiratory distress due to bronchiolitis.
  Arms: Intervention: 3% Hypertonic Saline
Procedure: Intervention: Salbutamol (Ventolin) — In this arm of the study, participants will receive nebulized Salbutamol, a bronchodilator commonly used in the management of bronchospasm associated with respiratory conditions, including bronchiolitis. The objective is to evaluate the effectiveness of Salbutamol in comparison to 3% hypertonic saline in improving the clinical outcomes of infants with bronchiolitis.
  Arms: Intervention: Salbutamol (Ventolin)

SUMMARY:
Bronchiolitis is a common lower respiratory tract infection that often leads to hospitalization in infants. The use of nebulized 3% hypertonic saline for treating bronchiolitis is being explored as an alternative to Salbutamol. In nebulizers, normal saline serves as a diluent, allowing water molecules or drugs to be inhaled into the lungs. However, there has been limited research on this topic, and no local trials have been conducted.

This study aims to compare the effectiveness of 3% hypertonic saline and Salbutamol in treating bronchiolitis. A randomized controlled trial will be conducted at the Department of Pediatric Medicine, Services Institute of Medical Sciences, Lahore, over one year, involving 100 infants divided into two groups: one receiving 3% hypertonic saline and the other receiving Salbutamol. The RDAI score will be evaluated before and during treatment to assess recovery time. Data will be collected using a proforma and analyzed with SPSS v25. The study aims to determine which treatment leads to faster symptom control and shorter hospital stays, with significance defined as a p-value ≤0.05. The findings will guide future treatment choices for infants with bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis, an infection of the lower respiratory tract, is one of the common reasons why the infants are hospitalized. The effectiveness of nebulized hypertonic saline (3%) in case of bronchiolitis is under discussion around the globe. With the use of normal saline as the diluent in nebulizers and the oxygen as vaporizer, the water molecules or drugs can be breathed through the mouth or nose and spread to the respiratory tract and lungs by the airflow. This is how, Salbutamol can be replaced by 3% hypertonic saline. However, a little work has been done in the past and no trials has yet been conducted at local setup. The objective of this study is to compare the efficacy of 3% hypertonic saline versus Salbutamol in the treatment of bronchiolitis. A Randomized controlled Trial will be conducted at Department of Pediatric Medicine, Services Institute of Medical Sciences Lahore, for a period of one year. A sample size of 100 cases; 50 in each group will be included through Nonprobability consecutive sampling and will be divided randomly into two groups. In group H, 3% hypertonic saline solution will be provided. In group V, Salbutamol will be taken. Before and on the treatment day, the RDAI score will be examined for evaluation. A complete recovery time will be noted. Data will be filled in a proforma for record. SPSS v25 software will be used for data analysis. Both groups will be compared simultaneously to take mean time to control symptoms by using independent samples t-test and RDAI score. P-value ≤0.05 will be taken as significant. Therefore, selecting an appropriate drug with less chances of failure can be proved fruitful and can significantly reduce the hospital stay with early recovery. The results of this study will help to choose a better drug in future in the treatment of infants against bronchiolitis

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 2-24 months
* Gender; Both Male and female patients.
* Presenting with bronchiolitis (as per operational definition)

Exclusion Criteria:

Infant with metabolic disorder

* Congenital heart disease
* Immune deficiency

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-02-06 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in Respiratory Distress Assessment Instrument (RDAI) Score | 5 days
  The outcome measures of this study include the change in Respiratory Distress Assessment Instrument , assessed at baseline and on days 1, 2, 3, 4, and 5 of treatment, as well as the time to complete recovery, defined as achieving an score of less than 5.

IPD SHARING:
Plan to Share IPD: No